CLINICAL TRIAL: NCT02928627
Title: Hepatic and Circulating microRNAs miR-221 and miR-222 Expression and Its Clinical Significance in Hepatocellular Carcinoma (HCC)
Brief Title: Clinical Significance of Hepatic and Circulating microRNAs miR-221 and miR-222 in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: Robert Gordon University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-035-16
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2016-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * hepatic tissue (matched tumoral/non tumoral) from patients with HCC
  * blood sample from patients with HCC and from healthy controls
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCC Group: samples obtained from patients with HCC (hepatic tissue and blood)
  Interventions: Other: Analysis of microRNA expression
- Plasma control Group (PCG): blood samples obtained from healthy controls
  Interventions: Other: Analysis of microRNA expression

INTERVENTIONS:
Other: Analysis of microRNA expression — sample analysis

SUMMARY:
Hepatocellular carcinoma (HCC) is the most frequent primary tumour of the liver and is the third cause of cancer-related mortality worldwide. Depending on the stage of the disease, the treatment options are surgery, liver transplantation, chemotherapy or radiotherapy.

Recently, scientific research has focused on small molecules called microRNAs which are produced by human cells and can be released in the blood. They have a role in cell proliferation and are found to be dysregulated in different types of cancer.

It has been shown that microRNAs have a role in the development of HCC but it is unknown if these molecules can be used as markers for diagnosis and survival in HCC.

In particular, microRNAs miR-221 and miR-222 are dysregulated in the tumoral tissues in about 80% of patients with HCC. This can be assessed on tissues from liver biopsies or surgical specimens, both invasive approaches. Only few studies showed the presence of microRNAs in the blood of patients with HCC but it is unknown if there is a correlation between tumoral tissue expression and circulating levels.

The aim of this study is to evaluate if these two microRNAs are expressed not only in the tumoral tissues but also in the blood from cancer patients, and in different amounts compared to circulating levels in healthy individuals. A correlation between tumoral tissue and blood levels will also be evaluated.

Should this evaluation show a strong correlation and reliability of circulating microRNAs in the diagnosis and follow up of HCC, future clinical trials targeting these microRNAs and their related pathways might benefit from this being adopted as conventional practice instead of the need of assessing tissue levels from liver biopsies.

The results of this pilot study will bring preliminary results as a first step for future analysis on a larger cohort of patients.

DETAILED DESCRIPTION:
1. Background & Rationale Hepatocellular carcinoma (HCC) is the sixth most prevalent cancer worldwide, and is the third cause of cancer-related mortality.

   Surgical resection remains the best curative treatment option for patients with clinical Barcelona-Clinic Liver Cancer (BCLC) stage A disease and it has shown benefits even in the more advanced stage B with multifocal disease or limited vascular invasion.

   Despite curative treatments offering a 5-year survival rate of 50-70%, recurrence rates at 5 years after surgery are as high as 70%. Therefore, more efforts are needed in order to identify prognostic factors for recurrence and survival.

   MicroRNAs are a class of small non-coding RNAs molecules, which act as key regulators of cell proliferation, differentiation, apoptosis and embryonic development, finely tuning gene expression at post-transcriptional level. They act as oncogenes or tumor suppressors depending on the target genes. In HCC, it has been reported the upregulation or downregulation of a few cluster of microRNAs, with a subsequent activation of molecular networks such as b-catenin, Ras, TGF-b, JAK/STAT and creation of a highly controlled feedback mechanism.

   Their involvement in carcinogenesis represents an important area of investigation for the development of their clinical applications: diagnostics, monitoring and therapeutics. MicroRNA profiles can distinguish between normal and cancerous tissue, identify tissue of origin and also discriminate different subtypes or specific oncogenic abnormalities. Indeed, microRNA mis-expression patterns are more accurate in identifying the origin of tumours that are otherwise difficult to be determined, suggesting that tumours more clearly maintain a unique tissue microRNA expression profile.

   MicroRNAs could also be useful as early diagnosis biomarkers for patient follow-up.

   In liver tumorigenesis, the role of miR-221 and miR-222 has not been completely elucidated. Previous studies showed that miR-221 was upregulated in 83% of HCC tumoral samples when compared with matched cirrhotic tissue.

   Increased expression of serum miR-221 was found in HCC patients compared to healthy normal controls, which was associated with the presence of other poor prognostic factors and with poorer outcomes after liver resection.

   The extraction of microRNAs from liver samples is limited by the ability to resecting the tumour or the possibility to perform a liver biopsy in each patient. On the contrary, a blood sample is easy to be collected and stored for analysis. At present, it has not been clearly established a correlation between the expression of miR-221 and miR-222 in the liver tissue (tumoral and non tumoral) and the circulating miR-221 and miR-222 levels.

   The confirmation of this correlation, would allow identifying a cutoff of circulating levels which could be used as a surrogate marker in order to include HCC patients in phase 3 trials without the need for a liver biopsy, which is often contraindicated for clinical reasons and according to guidelines.

   This is a pilot study to evaluate the correlation between the overexpression of miR-221 and miR-222 in paired tumoral/non tumoral liver tissue and blood samples in patients with HCC and to identify a cutoff for the circulating levels to use as a surrogate marker in clinical trials.

   This study therefore aims to evaluate if miR-221 and miR-222 expression in the blood correlates with tissue expression and if the circulating levels could be used as a surrogate of overexpression in the tumoral liver tissue.

   Should this evaluation show a strong correlation and reliability of circulating miRNAs, in the diagnosis and follow up of HCC, future clinical trials targeting these miRNAs and their related pathways might benefit from this being adopted as conventional practice instead of the need of assessing tissue levels from liver biopsies.

   The trial will be conducted in compliance with the principles of the Declaration of Helsinki, the principles of GCP and all (if any) applicable regulatory requirements are essential.

   NHS Grampian Biorepository will provide the anonymised samples to be used for this study. NHS Grampian Biorepository already has ethical approval in place for these types of studies. Research and Development approval will be sought.
2. Methods Blood samples from patients with HCC and from age-matched healthy controls, stored in the National bio-repository Scotland, will be tested for circulating miR-221 and miR-222 expression by the means of Real Time Reverse Transcription Polymerase Chain Reaction (RT-qPCR). Similarly, levels of miR-221 and miR-222 will be assessed in paired cancer and healthy liver tissue form patients with HCC.

   Sample analysis will take place in the Institute for Health and Wellbeing Research laboratory at Robert Gordon University (RGU) - Aberdeen.

   Results from the analysis of samples and quantification of microRNAs via RT-qPCR will be carried out by the chief investigator along with the research team in the laboratory facilities.

   Samples will be analysed to assess miR-221 and miR-222 overexpression between tumoral and non tumoral liver tissue and to assess the correlation between this and circulating miR-221 and miR-222. Circulating levels will be compared to results from age-matched healthy controls.

   The custodian of the data generated by the study will be the Chief Investigator.

   Samples will be stored in the laboratory facilities at RGU and only the chief investigator and the research team will have access to.

   Data generated by the study will be collected in a spreadsheet which will be bespoke and held on the intranet with access restricted only to the CI and the research team.

   Anonymised data on computer files will be stored on password-protected databases accessible only to the study investigators.

   All written files will be stored in locked filling cabinets within a secure store at Robert Gordon University with the exception of consents which are stored by NHS Grampian Biorepository.

   The University of Aberdeen and NHS Grampian monitoring procedures will be followed.

   At the end of the research the samples will be stored by research team pending ethical approval for use in another project, whereas the data generated by the study will be stored on password-protected databases accessible only to the study investigators.
3. Consent Process NHS Grampian Biorepository seek informed consent by patients for collection of tissue samples and blood through a dedicated research nurse and the use of a patient information sheet and a consent form which are part of the NHS Grampian Biorepository documentation.

   A consent will be obtained for all the samples used in this study according to the Biorepository consent process.
4. Trial Flowchart

   * Five frozen paired hepatic tumoral and non tumoral tissue and five frozen plasma samples obtained from patients with HCC and stored in the National Bio-Repository Scotland (HCC Group, HCC). Five voluntary age-matched healthy controls will be recruited to relate the expression of circulating miRNAs (Plasma Control Group, PCG).
   * Paired frozen HCC tissue specimens and their adjacent non-cancerous normal liver will be collected in RNA Stabilisation tubes and stored at -80C until further analysis and miRNAs extraction as per protocol. The average size of the specimen will be 2 by 10 mm in diameter.
   * Blood samples collected from both HCC Group and PCG (8-10ml, into BD Vacutainer K3-EDTA blood collection tubes) will be collected. All samples will be sent to Bio-Repository for further processing and then analysis and miRNAs extraction as per protocol.
   * The results of miRNAs extraction from paired HCC/non-cancerous tissues will be compared and from HCC Group plasma will be compared to the matched plasma of controls (PCG Group).

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma, not eligible for liver transplant undergoing surgical resection

Exclusion Criteria:

* extrahepatic disease, other primary tumour

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient affected by hepatocellular carcinoma undergoing curative surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-10 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
presence of miR-221 and mR-222 in the blood | 6 months
  To evaluate the presence of miR-221 and mR-222 in the blood of patients with HCC compared to age-matched healthy controls

SECONDARY OUTCOMES:
correlation of expression of miR-221 and miR-222 in tissue and blood samples | 6 months
  To evaluate the correlation between the expression of miR-221 and miR-222 in tissue and blood samples in patients with HCC

CONTACTS AND LOCATIONS:
Overall Officials: Fiammetta Soggiu, MD, Principal Investigator — NHS Grampian
Locations (1):
- Fiammetta Soggiu, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qi J, Wang J, Katayama H, Sen S, Liu SM. Circulating microRNAs (cmiRNAs) as novel potential biomarkers for hepatocellular carcinoma. Neoplasma. 2013;60(2):135-42. doi: 10.4149/neo_2013_018. PMID 23259781
- [Background] Gramantieri L, Ferracin M, Fornari F, Veronese A, Sabbioni S, Liu CG, Calin GA, Giovannini C, Ferrazzi E, Grazi GL, Croce CM, Bolondi L, Negrini M. Cyclin G1 is a target of miR-122a, a microRNA frequently down-regulated in human hepatocellular carcinoma. Cancer Res. 2007 Jul 1;67(13):6092-9. doi: 10.1158/0008-5472.CAN-06-4607. PMID 17616664
- [Background] Li J, Wang Y, Yu W, Chen J, Luo J. Expression of serum miR-221 in human hepatocellular carcinoma and its prognostic significance. Biochem Biophys Res Commun. 2011 Mar 4;406(1):70-3. doi: 10.1016/j.bbrc.2011.01.111. Epub 2011 Feb 3. PMID 21295551